CLINICAL TRIAL: NCT01122368
Title: An Exploratory Study to Compare the Efficacy and Safety of Micafungin as a Pre-emptive Treatment of Invasive Candidiasis Versus Placebo in High Risk Surgical Subjects - A Multicentre, Randomized, Double-blind Study
Brief Title: A Study to Evaluate Pre-emptive Treatment for Invasive Candidiasis in High Risk Surgical Subjects
Acronym: INTENSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 9463-EC-0002; 2008-006409-18 (EudraCT Number)
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Mycoses
Keywords: mycoses; Micafungin; intra-abdominal surgery; invasive fungal infection; intra-abdominal infection
MeSH Terms: conditions — Mycoses; Invasive Fungal Infections; Intraabdominal Infections | interventions — Micafungin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Micafungin (Experimental): IV
  Interventions: Drug: micafungin
- 2 Placebo (Placebo Comparator): IV
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: micafungin — IV
  Other Names: FK463; mycamine
  Arms: 1 Micafungin
Drug: placebo — IV
  Arms: 2 Placebo

SUMMARY:
Subjects with intra-abdominal infection requiring surgery and Intensive Care Unit stay will be treated early with micafungin or placebo to determine the incidence and time to confirmation of fungal infection.

DETAILED DESCRIPTION:
Subjects will be assessed at the following visits:

* Baseline (after surgery, prior to randomization)
* End of Treatment (EOT) visit (EOT is defined as: requires alternative antifungal, sufficient improvement of surgical condition, confirmed fungal infection or death)
* End of Study visit (28 days after the EOT visit)
* Long-term Follow up visit (90 days after the EOT visit)

ELIGIBILITY:
Inclusion Criteria:

* Intra-abdominal infection requiring surgery and Intensive Care Unit stay
* If Community Acquired Intra-Abdominal Infection, at least 72 hours (but not more than 120 hours) of Intensive Care Unit stay, counted from the end of surgery, and a further expected duration of Intensive Care Unit stay of ≥ 48 hours
* If Nosocomial Intra-Abdominal Infection, duration of Intensive Care Unit stay ≤ 48 hours, counted from the end of surgery, and a further expected duration of Intensive Care Unit stay of ≥ 48 hours
* Female subject of childbearing potential must have a negative urine or serum pregnancy test prior to randomization and must agree to maintain highly effective birth control during the study

Exclusion Criteria:

* Acute pancreatitis
* Neutropenia (ANC <1,000/mm3) at the time of randomization
* Infected intra-peritoneal dialysis
* Patients undergoing solid organ transplantation
* Documented invasive candidiasis at the time of randomization
* Expected survival < 48 hours
* Any systemically active anti-fungal within 14 days prior to administration of the study drug
* Allergy, hypersensitivity, or any serious reaction to an echinocandin anti-fungal or any of the study drug excipients
* Currently receiving and/or has taken an investigational drug within 28 days prior to randomization
* Pregnant woman or breast-feeding mother
* 'Do Not Resuscitate' order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2010-07-13 (Actual); Primary Completion 2011-12-15 (Actual); Study Completion 2011-12-15 (Actual)

PRIMARY OUTCOMES:
The incidence of Invasive Fungal Infection | During treatment
Time from baseline to the first confirmation of Invasive Fungal Infection | Baseline to End of Treatment visit

SECONDARY OUTCOMES:
The incidence during the treatment period and the time to confirmation of the composite endpoint (defined as confirmation of Invasive Fungal Infection and/or administration of alternative anti-fungal therapy) | At the EOT visit
The emergence or persistence of fungal colonization | At the EOT visit
The level of organ dysfunction | At the EOT visit
To assess the requirement for additional abdominal surgery/intervention. | At the End of Study visit
Organ failure-free days | From Day 1 until 28 days after end of study drug treatment
Fungal-free survival | From Day 1 until 28 days after end of study drug treatment
Intensive Care Unit (ICU)-free days | From Day 1 until 28 days after end of study drug treatment
All-cause mortality | At the End of Study and Long-Term Follow Up visit
Health-related quality of life | At the End of Study visit
Assessment of the safety of micafungin when used as a pre-emptive treatment | At the End of Study visit

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe Ltd.
Locations (49):
- Austria (3):
  - Innsbruck
  - Salzburg
  - Vienna
- Belgium (4):
  - Brussels
  - Edegem
  - Ghent
  - Liège
- Viborg, Denmark
- Finland (3):
  - Jyväskylä
  - Kuopio
  - Tampere
- France (6):
  - Amiens
  - La Roche-sur-Yon
  - Limoges
  - Paris
  - Pierre-Bénite
  - Poitiers
- Germany (5):
  - Cologne
  - Freiburg im Breisgau
  - Hanover
  - Leipzig
  - Lübeck
- Greece (2):
  - Athens
  - Thessaloniki
- Hungary (3):
  - Debrecen
  - Győr
  - Szeged
- Israel (2):
  - Ramat Gan
  - Tel Aviv
- Italy (6):
  - Bologna
  - Milan
  - Monza
  - Pisa
  - Roma
  - Verona
- Romania (3):
  - Bucharest
  - Oradea
  - Timișoara
- Spain (4):
  - Barcelona
  - Madrid
  - Valencia
  - Valladolid
- Lausanne, Switzerland
- Turkey (Türkiye) (4):
  - Ankara
  - Ege
  - Eskişehir
  - Trabzon
- United Kingdom (2):
  - Blackpool
  - Leeds

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] White PL, Posso R, Parr C, Price JS, Finkelman M, Barnes RA. The Presence of (1-->3)-beta-D-Glucan as Prognostic Marker in Patients After Major Abdominal Surgery. Clin Infect Dis. 2021 Oct 5;73(7):e1415-e1422. doi: 10.1093/cid/ciaa1370. PMID 32914187
- [Derived] Knitsch W, Vincent JL, Utzolino S, Francois B, Dinya T, Dimopoulos G, Ozgunes I, Valia JC, Eggimann P, Leon C, Montravers P, Phillips S, Tweddle L, Karas A, Brown M, Cornely OA. A randomized, placebo-controlled trial of preemptive antifungal therapy for the prevention of invasive candidiasis following gastrointestinal surgery for intra-abdominal infections. Clin Infect Dis. 2015 Dec 1;61(11):1671-8. doi: 10.1093/cid/civ707. Epub 2015 Aug 13. PMID 26270686
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=211